CLINICAL TRIAL: NCT00571805
Title: Placebo-controlled Study of Varenicline Effects on Nicotine Withdrawal Followed by a Test of Smoking Topography, Reward, and Reinforcement
Brief Title: Study of Varencline Effects on Cigarette Smoking Reward and Craving During a Model of Brief Quit Attempt
Acronym: VarenSmoke
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Malcolm S. Reid, PhD, New York University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Varenicline/Smoking; GA30513U
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Nicotine Dependence
Keywords: cigarette; craving; reward
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Varenicline
  Interventions: Drug: varencline
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varencline — 2.0 mg/day varencline (1.0 mg BID)
  Other Names: Chantix
  Arms: 1
Drug: placebo — matching placebo
  Arms: 2

SUMMARY:
Study of varenicline 2.0 mg/day treatment for 2 weeks with smoking test done in laboratory on Day 8 and a 1 week quit attempt from Day 8-14.

ELIGIBILITY:
Inclusion Criteria:

* At least 10 cigarettes/day
* Interest in quitting smoking
* Willgness to comply with overnight smoking abbstiennce period followed by lab smoking test

Exclusion Criteria:

* Pregnancy
* Axis I psychiatric disorder which require treatment with psychoactive medication and would make study compliance difficult.
* Clinically significant medical condition in opinion of study clinician
* Drug or alcohol dependence inlast 12 months
* Use of other smoking cessation medications ot treatment progams in last 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09

PRIMARY OUTCOMES:
Smoking reward | laboratory test

SECONDARY OUTCOMES:
1 week abstinence induced craving and reward | Day 8, 9, 11 and 14 questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Reid, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- VA New York Harbor Healthcare System, MHAD clinic, New York, New York, United States